CLINICAL TRIAL: NCT07263997
Title: Assessment of a New Traction Device in Submucosal Dissection of Colorectal Lesions
Acronym: COLOTRACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A01865-44
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer (MSI-H)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SureTrac aArm (Experimental): SureTrac™ traction device i sused to perform submucosal dissection
  Interventions: Device: SureTrac is designed to perform single or multi-polar traction and to adjust the traction intensity during dissection.

INTERVENTIONS:
Device: SureTrac is designed to perform single or multi-polar traction and to adjust the traction intensity during dissection. — The SureTrac device consists of a main attachment clip to which an elastic silicone device comprising four aligned rings is attached. The device is designed to retract and release elastic potential energy for dynamic traction. This allows for better visualisation of tissues and facilitates Submucosal dissection of colorectal lesions.

SUMMARY:
Colorectal cancer is a major public health issue. In France, in 2015, there were 40,000 new cases and 17,000 deaths. It develops from adenomas or scalloped polyps, which are usually accessible for endoscopic resection.

Piece-meal mucosectomy is the standard technique in Europe and the USA for lesions larger than 2 cm. It has certain advantages, such as its ease of learning, low morbidity and speed of execution. However, it has one major disadvantage, namely the low rate of monobloc resection and R0 for lesions larger than 2 cm.

Submucosal dissection (SMD) has become the standard technique for endoscopic resection of superficial colorectal lesions larger than 2 cm, particularly if the lesion presents a risk of superficial degeneration. Unlike mucosectomy, this technique allows for monobloc resection targeting R0 for all types of superficial lesions without size limitations, enabling histological analysis without data loss and with a recurrence rate of less than 2%.

However, there are numerous disadvantages to dissection:

* SMD is more difficult than mucosectomy, with a long learning curve, limiting its use to expert centres.
* The morbidity of dissection is higher than that of mucosectomy, with a risk of perforation of 4% vs. 1%.
* The procedure takes on average three times longer than mucosectomy.

From a technical standpoint, various methods have been described to facilitate the procedure, in particular traction using clips and elastic bands, which is the most widely used method in France.

Micro-Tech offers a new traction device, SureTrac, which is designed to perform single or multi-polar traction and to adjust the intensity of traction during dissection. The product is CE marked but has not yet been distributed in France. No data are currently available in the literature on this product other than a case report submitted for publication. A pilot study conducted by an expert centre is therefore necessary. This is why this study is being initiated.

DETAILED DESCRIPTION:
Colorectal cancer is a major public health issue. In France, in 2015, there were 40,000 new cases and 17,000 deaths. It develops from adenomas or scalloped polyps, which are usually accessible for endoscopic resection.

The larger the size of the colonic lesion, the higher the risk of degeneration, and the more difficult and risky endoscopic resection becomes. Nevertheless, this risk is still lower than that of surgery, which has a morbidity rate of 24%.

Piece-meal mucosectomy is the standard technique in Europe and the USA for lesions larger than 2 cm. It has certain advantages, such as its ease of learning, low morbidity and speed of execution. However, it has one major disadvantage, namely the low rate of monobloc resection and R0 for lesions larger than 2 cm. In this indication, it is therefore debatable because the risk of recurrence is 15%, or even 30% for lesions larger than 4 cm. Histological analysis is potentially less reliable, with the risk of losing histological fragments and only partially examining the specimens. This can potentially bias the decision to perform additional surgery or follow-up. Finally, the need to perform repeated colonoscopies in the event of recurrence or during monitoring leads to additional costs and a loss of patient follow-up.

Submucosal dissection (SMD) has become the standard technique for endoscopic resection of superficial colorectal lesions larger than 2 cm, particularly if the lesion presents a risk of superficial degeneration. Unlike mucosectomy, this technique allows for monobloc resection targeting R0 for all types of superficial lesions without size limitations, enabling histological analysis without data loss and with a recurrence rate of less than 2%.

However, there are numerous disadvantages to dissection:

* SMD is more difficult than mucosectomy, with a long learning curve, limiting its use to expert centres.
* The morbidity of dissection is higher than that of mucosectomy, with a risk of perforation of 4% vs. 1%.
* The procedure takes on average three times longer than mucosectomy.

From a technical standpoint, various methods have been described to facilitate the procedure, in particular traction using clips and elastic bands, which is the most widely used method in France. This involves pulling the lesion using a clip and elastic band to open up the submucosal layer and facilitate dissection. Certain variations have been described, such as multi-traction and adaptive traction, which are performed using non-dedicated, off-label devices (haemostatic clip and dental elastic band).

Micro-Tech offers a new traction device, SureTrac, which is designed to perform single or multi-polar traction and to adjust the intensity of traction during dissection. The product is CE marked but has not yet been distributed in France. No data are currently available in the literature on this product other than a case report submitted for publication. A pilot study conducted by an expert centre is therefore necessary. This is why this study is being initiated.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years old
* Patient with a colorectal lesion larger than 2 cm
* Patient eligible for SMD with elastic traction
* Patient affiliated with or beneficiary of a social security scheme
* French-speaking patient who has signed an informed consent form

Exclusion Criteria:

* Patients in poor general health who should not undergo endoscopy.
* Patients with an upper digestive tract that cannot be accessed by the endoscope.
* Patients with severe coagulation disorders and diseases associated with a risk of haemorrhage (platelets <50G/L, PT < 50%, INR > 1.5, APTT >1.5).
* Patients who are allergic to the instrument and to the drugs administered during the operation
* Patients who are not compatible with the use of the product according to the diagnosis Patients with lesions located in the appendix, ileocecal valve or within a diverticulum
* Patients with lesions that present a risk of deep submucosal invasion based on their morphological appearance (Kudo lesion > 10 mm or Sano IIIB > 10 mm or connect III)
* Patients with recurrence of a lesion previously resected by endoscopy or surgery
* Patients with a history of chronic inflammatory bowel disease (IBD) or familial adenomatous polyposis (FAP)
* Patients with a history of pelvic radiotherapy
* Patients for whom follow-up data cannot be collected
* Pregnant women
* Protected patients: adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision
* Patients hospitalised without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Submucosal dissection feasibility with the SureTrac traction device. | Day 0 (resection day)
  Feasibilty will be the rate of monobloc resection with the SureTrac device. Monobloc resection requiring another device or fragmented resection (regardless of the device) will be considered a failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No